CLINICAL TRIAL: NCT02669485
Title: A Prospective Study to Investigate the Impact of Using Indocyanine Green-enhanced Fluorescence Imaging on the Location of Bowel Transection in Patients Undergoing Left-sided Colorectal Resection
Brief Title: The Impact of Indocyanine Green-enhanced Fluorescence Imaging on Bowel Transection in Left-sided Colorectal Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Dominic C.C. Foo, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UW 16027
Record Dates: First submitted 2016-01-21; First posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Anastomotic Leak
Keywords: ICG; colectomy; anastomotic leak; anastomotic leakage rate; surgical decision
MeSH Terms: conditions — Anastomotic Leak | interventions — Indocyanine Green; Optical Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ICG (Experimental): Administering indocyanine green during surgery and the use of ICG fluorescence imaging to assess bowel perfusion during surgery
  Interventions: Drug: indocyanine green; Device: Fluorescence imaging

INTERVENTIONS:
Drug: indocyanine green — Injection of indocyanine green and using fluorescence imaging to assess perfusion of bowel before bowel transection and anastomosis
Device: Fluorescence imaging

SUMMARY:
The aim of this study was to evaluate the impact of fluorescence imaging on the location of colorectal transection lines based on evaluation of perfusion with indocyanine green, how it's going to affect surgical planning and its possible benefits in reducing anastomotic leakage.

DETAILED DESCRIPTION:
During surgery, the line of intended bowel transection would be determined by the surgeon. Then the anesthesiologist will administer a bolus of 5mg ICG intravenously (2.5mg/ml, 2ml), followed by 10ml normal saline flush. The perfusion of colon will be assessed via fluorescence angiography. The actual bowel transection, after ICG fluorescence study, would be compared with the intended bowel transection site. The difference in terms of distance and either more proximal or distal is recorded. Then bowel anastomosis is completed in the usual manner.

ELIGIBILITY:
Inclusion Criteria:

* All left-sided colorectal resection involving division of inferior mesenteric artery

Exclusion Criteria:

* Patients with a history of adverse reaction or known allergy to ICG, iodine, or iodine dyes. Pregnant and/or lactating patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with operative decisions changed after the use of ICG enhanced fluorescence imaging | intraoperative

SECONDARY OUTCOMES:
Anastomotic leak | up to 2 weeks after operation

CONTACTS AND LOCATIONS:
Overall Officials: Dominic, Chi Chung Foo, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JC, Lee JL, Yoon YS, Alotaibi AM, Kim J. Utility of indocyanine-green fluorescent imaging during robot-assisted sphincter-saving surgery on rectal cancer patients. Int J Med Robot. 2016 Dec;12(4):710-717. doi: 10.1002/rcs.1710. Epub 2015 Oct 21. PMID 26486376
- [Background] Hellan M, Spinoglio G, Pigazzi A, Lagares-Garcia JA. The influence of fluorescence imaging on the location of bowel transection during robotic left-sided colorectal surgery. Surg Endosc. 2014 May;28(5):1695-702. doi: 10.1007/s00464-013-3377-6. Epub 2014 Jan 3. PMID 24385249
- [Background] Jafari MD, Wexner SD, Martz JE, McLemore EC, Margolin DA, Sherwinter DA, Lee SW, Senagore AJ, Phelan MJ, Stamos MJ. Perfusion assessment in laparoscopic left-sided/anterior resection (PILLAR II): a multi-institutional study. J Am Coll Surg. 2015 Jan;220(1):82-92.e1. doi: 10.1016/j.jamcollsurg.2014.09.015. Epub 2014 Sep 28. PMID 25451666
- [Background] Gurtner GC, Jones GE, Neligan PC, Newman MI, Phillips BT, Sacks JM, Zenn MR. Intraoperative laser angiography using the SPY system: review of the literature and recommendations for use. Ann Surg Innov Res. 2013 Jan 7;7(1):1. doi: 10.1186/1750-1164-7-1. PMID 23289664